CLINICAL TRIAL: NCT05812898
Title: Effects of Adding Deep Front Line Myofascial Release to Selected Exercises in Patients With Knee Osteoarthritis
Brief Title: Adding Deep Front Line Myofascial Release to Selected Exercises in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hoda mohamed Ahmed, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004281
Record Dates: First submitted 2023-04-01; First posted 2023-04-14 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Knee Osteoarthritis
Keywords: myofascial release; Knee osteoarthritis; Deep front line
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise; Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: exercise plus myofascial release of the adductor and tipialis posterior muscles.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Sham Comparator): The control group received selective exercises therapy in the form of strengthening and stretching exercises for selective muscles of hip and knee
  Interventions: Other: exercises
- study group (Experimental): The study group received selective exercises therapy in the form of strengthening and stretching exercises for selective muscles of hip and knee, plus myofascial release technique of the deep front line.
  Interventions: Other: exercises; Other: myofascial release

INTERVENTIONS:
Other: exercises — strengthening of the gluteus maximus and medius, calf muscles stretching for calf and hamstring muscles
Other: myofascial release — myofascial release using instrument assisted soft tissue mobilization
  Arms: study group

SUMMARY:
the aim of the study is to investigate the effect of deep front line myofascial release to selected exercises in patients with knee osteoarthritis

DETAILED DESCRIPTION:
: Knee osteoarthritis (KOA) also known as degenerative joint disease, is typically the result of wear and tear and progressive loss of articular cartilage.

The myofascial meridian is a new approach to the facial restriction .the knee capsules, the adductor muscles and the tipialis posterior are part of the deep front line which is a line of the myofascial meridian.

Exercise is the highest evidence in the treatment of knee osteoarthritis. The myofascial release is effective in the treatment of knee osteoarthritis so the study will investigate the effect of adding deep front line myofascial release to selected exercises in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate unilateral or bilateral medial tibiofemoral OA grade II-III (K/L).
* The age of the participants will range from 45 to 60 years old .
* BMI ranged from 20-30 kg/m2

Exclusion Criteria:

1. Severe knee OA (grade IV according to K/L classification).
2. Congenital or acquired inflammatory, rheumatic or neurological (systemic or local) diseases involving the knee.
3. Patients receiving oral or injected corticosteroids for the last 3 months .
4. History of knee surgery/fracture.
5. Patients with ACL and meniscus injury

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  The scale that will be used the visual analogue scale;each subject will instructed to record pain intensity on line of 100mm. Starting from no pain on the leftto the most sever pain imaginable on the right Patient will choose the point which describe his pain.the more the score toward the end the more severe pain
function | up to four weeks
  The Arabic version of reduced Western Ontario and McMasters University Osteoarthritis Index (ArWOMAC) index will be used to measure functional disability.is a self-administered questionnaire consisting of 24 items divided into 3 subscales:
  * Pain (5 items): During walking, using stairs, in bed, sitting or lying, and standing upright
  * Stiffness (2 items): After first waking and later in the day Physical Function (17 items).The scores for each subscale are summed up, with a possible score range of 0-20 for Pain, 0-8 for Stiffness, and 0-68 for Physical Function.Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations
rang of motion | up to four weeks
  using digital inclinometer
joint position sense | up to four weeks
  using digital inclinometer for target angle 30 degree knee flexion

CONTACTS AND LOCATIONS:
Overall Officials: hoda m Ahmed, bachelor, Principal Investigator — phyical therapist at Cairo university hospitals
Locations (1):
- Hoda Mohamed Ahmed, Giza, Egypt